CLINICAL TRIAL: NCT00642538
Title: A Phase 1, Repeated Single-Dose, Double Blind, Randomized, Five Treatment Controlled Safety and Pharmacological Response Evaluation Trial of MKC253 Inhalation Powder in Adult Male and Postmenopausal Female Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study Designed to Determine the Safety and Pharmacological Response ofMKC253 Inhalation Powder in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MKC-253-002; EudraCT #: 2007-003430-42
Record Dates: First submitted 2008-03-03; First posted 2008-03-25 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetic adult male, diabetic postmenopausal women
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental): 1.5 mg dose of GLP-1 as MKC253 Inhalation Powder
  Interventions: Drug: MKC253 Inhalation Powder
- 2 (Experimental): 1.5 mg dose of GLP-1 as MKC253 Inhalation Powder
  Interventions: Drug: MKC253 Inhalation Powder
- 3 (Experimental): 1.5 mg dose of GLP-1 as MKC253 Inhalation Powder
  Interventions: Drug: MKC253 Inhalation Powder
- 4 (Placebo Comparator): TIP (placebo comparison)
  Interventions: Drug: Technosphere Inhalation Powder
- 5 (Active Comparator): 10 ug subcutaneous control
  Interventions: Drug: subcutaneous injection

INTERVENTIONS:
Drug: MKC253 Inhalation Powder — Inhalation Powder, prandial
  Arms: 1; 2; 3
Drug: Technosphere Inhalation Powder — Inhalation Powder, prandial
  Arms: 4
Drug: subcutaneous injection — 10µg Exenatide, prandial
  Arms: 5

SUMMARY:
20 eligible subjects will be enrolled into the treatment phase of the trial.

DETAILED DESCRIPTION:
Trial objectives are to determine the safety & pharmacological response of MKC253 Inhalation Powder.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking males and females between 18 and 70 years of age
* Body Mass Index (BMI) of < 32 kg/m2
* Diabetes managed on a stable regimen of diet and exercise within the preceding 8 weeks and/or metformin and/or a sulfonylurea or meglitinide or alpha glucosidase inhibitors, without any dose adjustments within the preceding 8 weeks. For subjects taking both metformin and sulfonylurea or meglitinide or alpha glucosidase inhibitor, one or both oral agents must be less than 1/2 the maximal allowable dose as cited in the product label.
* HbA1c = 6.2 to = 8.5%. Fasting C-peptide = 0.5 ng/mL. On the last 3 days of the washout period (Day -3, -2, and -1) subjects should have a FBG (finger stick) = 13.5 mmol/L.
* Normal pulmonary function and performance on pulmonary function tests
* Written Informed Consent
* Treatment with any type of anti-diabetic therapy other than metformin, sulfonylurea, meglitinide and alpha glucosidase inhibitors within the preceding 12 weeks [ie, thiazolidinediones (TZDs), dipeptyl peptidase inhibitors (DPP-IV), Symlin (pramlintide acetate) and or Byetta (exenatide)].

Exclusion Criteria:

* Exposure to any investigational medications or devices within the previous 90 days prior to trial entry or participation in another clinical trial while participating in this trial.
* Use of any prescription medication within 90 days prior to screening, other than allowed anti-diabetic therapy, that has not been approved by the PI and Sponsor. The use of alpha blockers, antihypertensives, proton pump inhibitors and cholesterol medication as co-medications is allowed throughout the study.
* Significant improvement in pre- to post-bronchodilator spirometry (defined as an increase of 12% AND 200 mL in either FVC OR FEV1).
* Serum creatinine above Upper Limit of Normal (ULN) as defined by the laboratory
* Any other condition which, in the opinion of the PI, makes the subject unsuitable for the clinical trial, or could limit the validity of the informed consent and/or impair the subject's ability to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
AUC 0-240 min post-prandial serum glucose | 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Anders Boss, Study Director — Mannkind Corporation
Locations (1):
- University Medical Centre Groningen, Zuidlaren, Netherlands